CLINICAL TRIAL: NCT06912620
Title: Efficacy of Alternative RUTFs for Treatment of Child Wasting and Prevention of Relapse
Brief Title: Alternative RUTFs for Treatment of Child Wasting
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: AFRICSante (Unknown); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-RUTF
Record Dates: First submitted 2025-03-19; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Severe Acute Malnutrition; Moderate Acute Malnutrition; Wasting
Keywords: Severe Acute Malnutrition; Moderate Acute Malnutrition; Wasting; Ready-to-use Therapeutic Foods; RUTFs; Wasting relapse; Plant-based RUTF; Dairy-free RUTF; Peanut-free RUTF
MeSH Terms: conditions — Severe Acute Malnutrition; Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The products will be provided in identical packaging and the participants, the care providers, the investigators, and outcomes assessors will be blinded to treatment assessment. However, the products may taste different and thus participants may know that they are receiving an alternative RUTF if they are familiar with the standard RUTF product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard RUTF (Active Comparator): This is the control arm of the trial, in which children will receive the standard RUTF product for treatment of acute malnutrition
  Interventions: Dietary Supplement: Standard RUTF
- Soy-based RUTF (Experimental): This is an interventional arm of the trial, in which children will receive an alternative formulation, a soy-based RUTF
  Interventions: Dietary Supplement: Soy-based RUTF
- Soy-maize-sorghum-based RUTF (Experimental): This is an interventional arm of the trial, in which children will receive an alternative formulation, a soy-maize-sorghum-based RUTF
  Interventions: Dietary Supplement: Soy-maize-sorghum-based RUTF

INTERVENTIONS:
Dietary Supplement: Soy-based RUTF — This alternative formulation of ready-to-use therapeutic foods (RUTFs) is a peanut-free formula that includes dairy (milk powder) with added crystalline amino acids
  Arms: Soy-based RUTF
Dietary Supplement: Soy-maize-sorghum-based RUTF — This alternative formulation of ready-to-use therapeutic foods (RUTFs) is a peanut-free and dairy-free formula with added crystalline amino acids
  Arms: Soy-maize-sorghum-based RUTF
Dietary Supplement: Standard RUTF — This is the control, the standard, currently used formulation of ready-to-use therapeutic foods (RUTFs), which contains dairy and peanut ingredients
  Arms: Standard RUTF

SUMMARY:
Acute malnutrition is the most life-threatening form of undernutrition. Moderate and severe acute malnutrition (MAM, SAM) are effectively treated with ready-to-use therapeutic foods (RUTFs) but there is a need to lower the cost of treatment and improve treatment regimens to reduce risk of relapse MAM/SAM episodes following recovery. The currently used standard formulation of RUTF contains peanuts and dairy, which pose problems due to their high cost, the need to import ingredients to the Global South (in the case of dairy), and risk of aflatoxin (in the case of peanuts). Before alternative formulations of RUTF can be recommended, however, there is the need for data on the efficacy of these formulations on recovery rates and to what extent recovery is sustainable. Sustainable recovery implies a lower rate of post-treatment relapse.

The study objectives are as follows: (1) To assess the non-inferiority of soy-maize-sorghum (SMS-) RUTF and soy-based (S-) RUTF on treatment recovery to standard RUTF; (2) To assess the superiority of SMS-RUTF and S- RUTF on post-recovery relapse compared to standard RUTF; (3) To assess the costs of a treatment course of SMS-RUTF, S-RUTF, and standard RUTF; (4) To assess the effect of SMS-RUTF and S-RUTF on microbiome composition and intestinal inflammation

The investigators will conduct a facility-based, individually randomized controlled trial with three arms allocated in a 1:1:1 allocation ratio in 30 health facilities (Centre de Santé et Promotion Sociale [CSPS]) in Burkina Faso. The investigators will randomize 1080 children with MAM and 1080 children with uncomplicated SAM 6-59 months of age to receive treatment with one of the following RUTFs: (1) standard of care, milk- and peanut-based RUTF (control group); (2) SMS-RUTF free of milk and peanuts and high in fiber (intervention 1); or (3) S-RUTF free of milk and peanuts (intervention 2). Children will be enrolled upon presentation to facilities for MAM or uncomplicated SAM treatment. Follow up visits will be weekly during treatment for SAM children and bi-weekly during treatment for MAM children, and monthly for 3 months following discharge from treatment. The primary study outcomes include, among others, anthropometric recovery at discharge (a non-inferiority analysis) and relapse to MAM or SAM within the 3 months following recovery (a superiority analysis). The investigators will employ an activity-based micro-costing approach to collect cost data on the direct and indirect medical costs, opportunity costs to caregivers, personnel, and overheads associated with outpatient MAM or SAM treatment. Fecal samples will be collected from children at a subset of facilities (5 facilities, ~60 children per treatment arm), at enrollment (initiation of treatment), discharge from treatment, and 3-months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-59 months
* MUAC < 12.5 cm, or WLZ/WHZ < -2
* Absence of clinical complications or nutritional edema
* Pass the appetite test
* Accompanied by caregiver or legal guardian
* Caregiver or legal guardian consents to participate

Exclusion Criteria:

* Acute malnutrition requiring hospitalization (presence of clinical complications, failure to pass the appetite test, or presence of bilateral pitting edema)
* Known allergy to any of the ingredients in the RUTF products
* Already enrolled in MAM or SAM treatment program
* Presence of physical abnormalities that make measurement of anthropometry impossible
* Caregiver has intention to move out of the study area within the next 6 months
* Children referred from in-patient facilities to continue in ambulatory care

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2160 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Anthropometric recovery | At discharge, which is up to 12 weeks after admission
  Weight-for-length z-score (WLZ) ≥ -2 and middle upper arm circumference (MUAC) ≥ 125 mm and absence of bilateral pitting edema for two consecutive visits
Default from treatment | During treatment, which is up to 12 weeks after admission
  Child is absent for two consecutive visits, declared a defaulter on the second visit
Relapse to wasting | Within 3 months post-discharge
  A new episode of wasting (defined as weight-for-length/height z-score [WLZ/WHZ] < -2 or middle upper arm circumference [MUAC] < 125 mm or presence of bilateral pitting edema) within the 3-month period following recovery from the index wasting episode, among children who recovered from their index episode
Transfer to inpatient treatment | During treatment, which is up to 12 weeks after admission
  Referral or admission to hospital for inpatient treatment during the treatment course
Weight gain | During treatment, which is up to 12 weeks after admission
  Change in child's weight (gram/kilogram/day) between weight on day of admission to treatment and day of discharge
Non-response to treatment | During treatment, which is up to 12 weeks after admission
  Any of the following criteria are met: Absence of weight gain after 5 weeks or at the third visit; weight loss for more than 4 weeks in the program or at the second visit; loss of more than 5% of body weight compared to admission weight at any time; or anthropometric recovery criteria not met after 3 months of follow-up in treatment
Adherence to treatment services | During treatment, which is up to 12 weeks after admission
  Caregiver attends the recommended schedule of visits and receive ready-to-use therapeutic foods (RUTF) supply
Length of stay | During treatment, which is up to 12 weeks after admission
  The number of days between the day the child is admitted to treatment and the day the child is determined to be recovered and thus discharged from treatment
Anthropometry | At discharge, which is up to 12 weeks after admission
  Weight-for-length/height z-score (WLZ/WHZ), middle upper arm circumference (MUAC), weight, height/length, length/height-for-age z-score (LAZ/HAZ) and weight-for-age z-score (WAZ)
Relapse to MAM | Within 3 months post-discharge
  A new episode of MAM (weight-for-length/height z-score [WLZ/WHZ] <-2 and ≥-3, or middle upper arm circumference [MUAC] <125 mm and ≥115 mm) within the 3-month period following recovery from the index wasting episode
Relapse to SAM | Within 3 months post-discharge
  A new episode of SAM (weight-for-length/height z-score [WLZ/WHZ] < -3 or middle upper arm circumference [MUAC] < 115 mm or presence of bilateral pitting edema) within the 3-month period following recovery from the index wasting episode
Anthropometry | At 3 months post-discharge
  Weight-for-length/height z-score (WLZ/WHZ), middle upper arm circumference (MUAC), weight, height/length, length/height-for-age z-score (LAZ/HAZ) and weight-for-age z-score (WAZ)
Hemoglobin | At discharge, which is up to 12 weeks after admission
  Hemoglobin concentration (grams/liter)
Hemoglobin | At 3 months post-discharge
  Hemoglobin concentration (grams/liter)

SECONDARY OUTCOMES:
Morbidity | During treatment, which is up to 12 weeks after admission
  Indication of morbidity (acute respiratory infections, diarrhea, fever, or malaria) on health center card
Anemia | At discharge, which is up to 12 weeks after admission
  Hemoglobin concentration < 105 gram/liter for children 6-23 months of age Hemoglobin concentration < 110 gram/liter for children 24-59 months of age
Anemia | At 3 months post-discharge
  Hemoglobin concentration < 110 gram/liter
Mortality | During treatment, which is up to 12 weeks after admission, or during the 3-month post-discharge follow up
  Child has deceased

CONTACTS AND LOCATIONS:
Overall Officials: Laeticia Toe, Principal Investigator — Institut de Recherche en Sciences de la Santé
Locations (1):
- Health centers localted in the region of Hauts-Bassins, Bobo-Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the International Food Policy Research Institute's policy on research data management and open access, at the time of publication of scientific articles presenting results, the fully anonymized databases will become a public good and will be made available to the scientific community, government, and partners.
Supporting Information: Study Protocol, SAP